CLINICAL TRIAL: NCT02538692
Title: Traditional Chinese Medicine Tong-Xie-Yao-Fang Granules for Diarrhea-predominant Irritable Bowel Syndrome: a Randomized Placebo-controlled Trial and a Mechanistic Study
Brief Title: Tong-Xie-Yao-Fang Granules for Diarrhea-predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 81373644
Record Dates: First submitted 2015-08-30; First posted 2015-09-02 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tong-Xie-Yao-Fang (Experimental): Tong-Xie-Yao-Fang is a classic formula of traditional Chinese medicine for IBS-D. It is composed of 4 herbs: Radix Paeoniae Alba, Ledebouriella seseloides Wolff, pericarpium citri reticulatae and Rhizoma Atractylodis Macrocephalae. The granules will be administrated for thrice daily at a dose of 15g per time. The total duration of treatment is 4 weeks.
  Interventions: Drug: Tong-Xie-Yao-Fang
- Placebo (Placebo Comparator): It is a placebo that made with similar appearance and taste as the Tong-Xie-Yao-Fang granules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tong-Xie-Yao-Fang — Tong-Xie-Yao-Fang is a traditional Chinese formula. It is used for diarrhea management.
  Other Names: Tongxieyaofang
  Arms: Tong-Xie-Yao-Fang
Drug: Placebo — The placebo is the same as Tong-Xie-Yao-Fang in appearance.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the efficacy and safety of a traditional Chinese medication Tong-Xie-Yao-Fang for patients with diarrhea-predominant irritable bowel Syndrome (IBS-D).

DETAILED DESCRIPTION:
Participants: The sample size of this trial is 118, to test an odds ratio of 3.5 at a significance of 0.05 and power of 0.8.

Intervention: Tong-Xie-Yao-Fang versus placebo Data collection: Standard operation procedure will be developed for how to interviewing the participants, how to use the IBS diary, how to enter the data into the electronic case report forms.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed as IBS according to the Rome III criteria;
* Diarrhea was present for at least 75% of the time;
* With a TCM differentiation as "liver stagnation and spleen defficiency"
* Had a colonoscopy within a year to rule out other bowel diseases.

Exclusion Criteria:

* Organic gastrointestinal disease, such as colorectal cancer, inflammatory bowel disease, advanced colonic polyp;
* Had gastrointestinal surgery within a year;
* Used durgs that affect gastrointestinal motility;
* Had psychological disorder;
* Serious disease in other system, which may bias the outcome measures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
the proportion of patients who had adequate relief of global IBS-D symptoms for at least 2 of the 4 weeks. | 4 weeks after initiation of treatment

SECONDARY OUTCOMES:
Stool frequency per week | baseline(week 0), week 4, week 8, week 12
An visual scale rating the degree of IBS-D symptoms | baseline(week 0), week 4, week 8, week 12
  The scale ranges from 0 to 10. The score 0 indicates the mildest degree, while the 10 indicates the most serious degree.
Proportion of adverse events | week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Teaching Hospital of Chengdu University of TCM, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Chen M, Tang TC, Wang Y, Shui J, Xiao XH, Lan X, Yu P, Zhang C, Wang SH, Yao J, Zheng H, Huang DQ. Randomised clinical trial: Tong-Xie-Yao-Fang granules versus placebo for patients with diarrhoea-predominant irritable bowel syndrome. Aliment Pharmacol Ther. 2018 Jul;48(2):160-168. doi: 10.1111/apt.14817. Epub 2018 Jun 1. PMID 29856472